CLINICAL TRIAL: NCT01921361
Title: The Effects of Dexmedetomidine on Peroperative Shivering Incidence Under Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, RESUL ALTUNTAS, MD, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B.30.2.ERC.0.01.00.01/27
Record Dates: First submitted 2013-08-03; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Shivering; Dexmedetomidine; Spinal anesthesia
MeSH Terms: conditions — Postoperative Complications | interventions — Levobupivacaine; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous (Active Comparator): Intrathecal (3 ml) 15 mg levobupivacaine + 0.3 ml 0.9% Sodium chloride and intravenous dexmedetomidine (dexmedetomidine diluted 1mcg/ml and than 1ml/kg/10 minutes and 0.5 ml/kg/hour infusion)
  Interventions: Drug: Levobupivacaine; Drug: Dexmedetomidine; Drug: sodium chloride
- Intrathecal (Active Comparator): Intrathecal (3 ml) 15 mg levobupivacaine + (0.3 ml) 3 mcg dexmedetomidine (dexmedetomidine diluted 10 mcg/ml) and intravenous 0.9% Sodium chloride (1ml/kg/10 minutes and 0.5 ml/kg/hour infusion)
  Interventions: Drug: Levobupivacaine; Drug: Dexmedetomidine; Drug: sodium chloride
- Control (Placebo Comparator): Intrathecal (3 ml) 15 mg levobupivacaine + 0.3 ml 0.9% Sodium chloride and intravenous 0.9% Sodium chloride (1ml/kg/10 minutes and 0.5 ml/kg/hour infusion).
  Interventions: Drug: Levobupivacaine; Drug: sodium chloride

INTERVENTIONS:
Drug: Levobupivacaine — Intrathecal 3ml (15 mg)
  Other Names: Chirocaine, 0.5%, 10 ml, Abbott
Drug: Dexmedetomidine — Intrathecal 3 microgram (diluted 1/10, 0.3 ml)
  Other Names: Precedex, 100 mcg/ml, Abbott
  Arms: Intravenous
Drug: Dexmedetomidine — Intravenous 1ml/kg/10 minutes and than 0.5 ml/kg/hour infusion (dexmedetomidine diluted 1 microgram/ml)
  Other Names: Precedex, 100 mcg/ml, Abbott
  Arms: Intrathecal
Drug: sodium chloride — Intravenous 1ml/kg/10 minutes and than 0.5 ml/kg/hour infusion in the control and intrathecal groups, intrathecal 0.3 ml in the control and intravenous groups.
  Other Names: 0.9 Sodium chloride

SUMMARY:
The purpose of this study to compare the efficacy of intravenous or intrathecal dexmedetomidine on the incidence of shivering on patients who scheduled spinal anesthesia for elective surgery.

DETAILED DESCRIPTION:
The design of the study includes three study groups done in random order. The groups are as follows: 1) Control group received 15 mg levobupivacaine intrathecally and intravenous 0.9% sodium chloride; 2) Intravenous group received 15 mg levobupivacaine intrathecally and intravenous dexmedetomidine (1mcg/kg/10min, 0.5mcg/kg/h infusion) ; 3) Intrathecal group received 15 mg levobupivacaine + 3 mcg dexmedetomidine intrathecally and intravenous 0.9% sodium chloride.

Throughout the study period,shivering scores, tympanic temperature were recorded, heart rate were measured continuously using an electrocardiogram; blood pressure was determined oscillometrically at 5 min intervals at the ankle. In case heart rate decreased by more than 30% of the baseline atropin received and blood pressure decreased 30% of the baseline effedrin received.

Side effects (bradycardia, hypotension, hypothermia, nausea and vomiting etc ) were recorded peroperatively in the operating room and postanesthetic care unit.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 y/o patients
* American Society of Anesthesiologists' physical status class I-II
* Scheduled for the spinal anesthesia

Exclusion Criteria:

* Patients who have the body temperature over 37.3 celsius degree
* Pregnants
* Known allergies to the study drugs
* Contraindication to spinal anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
shivering score | 1 day (From start of anaesthesia till discharge from the recovery room )

SECONDARY OUTCOMES:
blood pressure | 1 day (From start of anaesthesia till discharge from the recovery room )
  non invasive blood pressure measured
heart rate | 1 day (From start of anaesthesia till discharge from the recovery room )
core temperature | 1 day (From start of anaesthesia till discharge from the recovery room )
  lower than 36 celsius degree was accepted as hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Resul Altuntas, MD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)